CLINICAL TRIAL: NCT03867708
Title: Outcomes of Transcatheter Closure of Secundum Atrial Septal Defect Guided by Three-dimensional Transesophageal Echocardiography
Brief Title: Outcomes of Transcatheter ASD Closure Guided by 3D-TEE
Status: Withdrawn | Type: Observational
Why Stopped: No participants found
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Aboelkasem Ali Mousa, Assistant lecturer, Assiut University
Other Study IDs: ASD closure guided by 3D-TEE
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: ASD2(Secundum Atrial Septal Defect)
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with residual shunt: patient with residual left to right shunt detected by 2D-TTE at 6 month follow up after ASD device closure guided by 3D-TEE
  Interventions: Radiation: ASD device closure
- patients without residual shunt: patient without residual left to right shunt by 2D-TTE at 6 month follow up after ASD device closure guided by 3D-TEE
  Interventions: Radiation: ASD device closure

INTERVENTIONS:
Radiation: ASD device closure — transcatheter secundum ASD device closure

SUMMARY:
Atrial Septal Defect (ASD) is a common cardiac diagnosis among adults.Three-dimensional transesophageal echocardiography (3D-TEE) improve the visualization of ASD, its rims and surrounding structures and can be used for guidance during percutaneous transcatheter closure. Proper device size selection is important for success of ASD device closure. 3D-TEE can assess the ASD morphology, maximal diameter, area and determine the device size without balloon sizing during percutaneous closure.There are some adverse outcomes reported in previous studies following transcatheter secundum ASD closure as: residual shunt, new onset atrial fibrillation(AF) and mitral regurgitation(MR)deterioration . These adverse outcomes are responsible for morbidity and mortality following transcatheter ASD closure, so it is essential to study risk factors associated with these adverse outcomes in order to minimize their incidence.The investigators will study the role of 3D-TEE in proper device size selection, also the percentage and predictors of adverse outcomes after device closure guided by 3D-TEE.

DETAILED DESCRIPTION:
The investigators will include 80 patients in a prospective cohort study .

For all patients the following study tools will be done:

1. Written consent.
2. Detailed history including Age, sex, symptoms (NYHA class).
3. Clinical examination.
4. Electrocardiogram (ECG) (to detect baseline rhythm).
5. Two-dimensional transthoracic echocardiography (2D TTE):

   All patients will undergo 2D TTE before device closure to assess:
   * ASD (type, size, shunt direction).
   * Pulsed Doppler quantification of the pulmonary (Qp) to systemic (Qs) blood flow ratio
   * Right ventricle (RV) enlargement: RV linear dimensions are best measured from a RV-focused apical four-chamber view.
   * RV systolic function by :

     1. Tricuspid annular plane systolic excursion(TAPSE) ,
     2. 2D RV fractional area change (FAC)= 100 X [(end-diastolic area - end-systolic area)/end-diastolic area)].
   * Pulmonary artery systolic pressure (PASP).
   * Grade of MR by Color Doppler: The color Doppler jet area of MR and left atrial area at the time of midsystole will be measured by the area trace method in the apical 4-chamber view, and the ratio of MR jet area to left atrial area will be calculated. The grade of MR will be determined by the ratio, where 0% to 10%>> none/trivial, 10% to 20% >> mild, 20% to 40% >>moderate, and >40% >> severe.
   * Left ventricle (LV) systolic function by m-mode,
   * LV diastolic function :

     1. Pulsed wave (PW) Doppler of trans-mitral flow during diastole.
     2. Tissue Doppler imaging (TDI).
6. Three-dimensional transesophageal echocardiography (3D-TEE):

   All patients will undergo 3D-TEE before device closure of secundum ASD to assess:
   1. The number of defects.
   2. Defect size: The maximum dimension (length), minor dimension (width), and area by planimetry will be measured from the 3D en face view.
   3. ASD morphology will be categorized by the shape seen in the en face view. ASD will be defined as circular when the minor dimension is >75% of the maximum length. If the minor dimension is <75% of the maximum length ASD will be defined as having an oval shape. Asymmetric, irregularly shaped defects that are not elliptical will be defined as having a complex shape.
   4. The surrounding rims: aortic rim, atrioventricular (AV) rim, superior vena cava (SVC) rim, inferior vena cava (IVC) rim and posterior rim.

   According to recent study, the optimal ASD device size will be calculated as :

   Device size = 0.964 x 3Dmax - 2.622 x circular index +7.084 Where maximal ASD diameter on 3D-TEE (3Dmax) and the circular index is defined as the ratio of the maximal to minimal diameters on the 3D-TEE image.
7. Transcatheter secundum ASD device closure procedure:

   All patients suitable for device closure will undergo transcatheter device closure procedure in cath lab under general anesthesia. After venous access is gained following local anesthesia via the right femoral vein, the ASD is crossed using a Multipurpose catheter. The Multipurpose catheter is then exchanged for a device-specific delivery system. Its tip is placed into the left atrium. The left-sided disk is then deployed and gently pulled back against the atrial septum under fluoroscopic guidance in a left anterior oblique projection. To deploy the right atrial disc, tension is maintained on the delivery cable while the delivery sheath is further withdrawn.

   The whole procedure will be under fluoroscopic and 3D-TEE guidance. Device size that will be used in ASD closure according to the previously mentioned formula based on 3D-TEE measurements.
8. Follow up:

   * Clinical follow up for 24 hours to detect post-ASD closure acute heart failure.
   * 2D-TTE will be performed 24 hours post-procedure to visualize the device position and to look for residual shunting and MR grade using color Doppler.
   * Clinical follow up, ECG and 2D-TTE at 6-month follow up to detect new onset AF, residual shunt and MR deterioration.
9. After 6 months of device closure :

Patients will be divided into two groups according to occurrence of adverse outcomes (residual shunt , MR deterioration and new onset AF ) and the following predictors will be evaluated in each group and their influence on occurrence of these adverse outcomes:

Echocardiographic data:

* RV systolic function by TAPSE and FAC on 2D-TTE.
* LV systolic function by m-mode on 2D-TTE.
* LV diastolic function on 2D-TTE.
* Estimated PASP on 2D-TTE.
* ASD shape on 3D-TEE.
* ASD maximal diameter on 3D-TEE.
* ASD minimal diameter on 3D-TEE.
* ASD area on 3D-TEE.
* Size of implanted device.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suitable indication for ASD closure according to recent guidelines :

  1. Impaired functional capacity.
  2. Right atrial and/or RV enlargement.
  3. Left-to-right shunt with [Qp: Qs] ≥1.5:1.
  4. Paradoxical embolism.
* Patients with isolated secundum ASD with sufficient rims suitable for device closure.

Exclusion Criteria:

* Small ASD with Qp/Qs <1.5:1 or no signs of RV volume overload
* A single defect too large for closure (>38 mm)
* Multiple ASDs unsuitable for percutaneous closure.
* Anterior, posterior, superior, or inferior rim <5 mm.
* Abnormal pulmonary venous drainage.
* Associated structural heart disease requiring cardiac surgery.
* ASD with severe pulmonary arterial hypertension and bidirectional or right-to-left shunting.
* Intracardiac thrombi diagnosed by echocardiography.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with secundum atrial septal defect with suitable rims for transcatheter device closure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Detection of residual shunt, MR deterioration and new onset AF following 3D-TEE guided ASD closure | six months
  Detection of residual shunt and MR deterioration by 2D-TTE and new-onset AF by ECG at six month follow up after ASD device closure

SECONDARY OUTCOMES:
Clinical outcomes after six months | six months
  Detection of mortality , cerebrovascular stroke and heart failure after six months of ASD device closure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mousa, Principal Investigator — Assiut University

REFERENCES:
- [Background] Alnasser S, Lee D, Austin PC, Labos C, Osten M, Lightfoot DT, Kutty S, Shah A, Meier L, Benson L, Horlick E. Long term outcomes among adults post transcatheter atrial septal defect closure: Systematic review and meta-analysis. Int J Cardiol. 2018 Nov 1;270:126-132. doi: 10.1016/j.ijcard.2018.06.076. Epub 2018 Jul 12. PMID 30054146
- [Background] Villablanca PA, Briston DA, Rodes-Cabau J, Briceno DF, Rao G, Aljoudi M, Shah AM, Mohananey D, Gupta T, Makkiya M, Ramakrishna H, Garcia MJ, Pass RH, Peek G, Zaidi AN. Treatment options for the closure of secundum atrial septal defects: A systematic review and meta-analysis. Int J Cardiol. 2017 Aug 15;241:149-155. doi: 10.1016/j.ijcard.2017.03.073. Epub 2017 Mar 24. PMID 28390741
- [Background] Silvestry FE, Cohen MS, Armsby LB, Burkule NJ, Fleishman CE, Hijazi ZM, Lang RM, Rome JJ, Wang Y; American Society of Echocardiography; Society for Cardiac Angiography and Interventions. Guidelines for the Echocardiographic Assessment of Atrial Septal Defect and Patent Foramen Ovale: From the American Society of Echocardiography and Society for Cardiac Angiography and Interventions. J Am Soc Echocardiogr. 2015 Aug;28(8):910-58. doi: 10.1016/j.echo.2015.05.015. No abstract available. PMID 26239900
- [Background] Chessa M, Carminati M, Butera G, Bini RM, Drago M, Rosti L, Giamberti A, Pome G, Bossone E, Frigiola A. Early and late complications associated with transcatheter occlusion of secundum atrial septal defect. J Am Coll Cardiol. 2002 Mar 20;39(6):1061-5. doi: 10.1016/s0735-1097(02)01711-4. PMID 11897451
- [Background] Rao PS, Langhough R. Relationship of echocardiographic, shunt flow, and angiographic size to the stretched diameter of the atrial septal defect. Am Heart J. 1991 Aug;122(2):505-8. doi: 10.1016/0002-8703(91)91008-b. PMID 1858633
- [Background] Gupta SK, Sivasankaran S, Bijulal S, Tharakan JM, Harikrishnan S, Ajit K. Trans-catheter closure of atrial septal defect: Balloon sizing or no Balloon sizing - single centre experience. Ann Pediatr Cardiol. 2011 Jan;4(1):28-33. doi: 10.4103/0974-2069.79619. PMID 21677801
- [Background] Kong WK. The relation between atrial septal defect area, diameter and shape using balloon sizing and three-dimensional transoesophageal echocardiography during percutaneous closure using occlutech device. Journal of the American College of Cardiology. 2017;69(11 Supplement):1493.
- [Background] Scacciatella P, Marra S, Pullara A, Conrotto F, Marchetti M, Ferraro G, Pavani M, Biasco L, Bongiovanni D, Gaita F, Orzan F. Percutaneous closure of atrial septal defect in adults: very long-term clinical outcome and effects on aortic and mitral valve function. J Invasive Cardiol. 2015 Jan;27(1):65-9. PMID 25589703
- [Background] Akagi T, Fujii Y, Takaya Y, Takahashi S, et al. Clinical benefit of transcatheter closure for newly developed atrial fibrillation in adult patients with atrial septal defect. Journal of the American College of Cardiology. 2018;71(11):A549.
- [Background] Takaya Y, Kijima Y, Akagi T, Nakagawa K, Oe H, Taniguchi M, Sano S, Ito H. Fate of Mitral Regurgitation After Transcatheter Closure of Atrial Septal Defect in Adults. Am J Cardiol. 2015 Aug 1;116(3):458-62. doi: 10.1016/j.amjcard.2015.04.042. Epub 2015 May 7. PMID 26026868
- [Background] Stout KK, Daniels CJ, Aboulhosn JA, Bozkurt B, Broberg CS, Colman JM, Crumb SR, Dearani JA, Fuller S, Gurvitz M, Khairy P, Landzberg MJ, Saidi A, Valente AM, Van Hare GF. 2018 AHA/ACC Guideline for the Management of Adults With Congenital Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Apr 2;73(12):e81-e192. doi: 10.1016/j.jacc.2018.08.1029. Epub 2018 Aug 16. No abstract available. PMID 30121239
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Johri AM, Witzke C, Solis J, Palacios IF, Inglessis I, Picard MH, Passeri JJ. Real-time three-dimensional transesophageal echocardiography in patients with secundum atrial septal defects: outcomes following transcatheter closure. J Am Soc Echocardiogr. 2011 Apr;24(4):431-7. doi: 10.1016/j.echo.2010.12.011. Epub 2011 Jan 22. PMID 21262563
- [Background] Jang JY, Heo R, Cho MS, Bae J, Hong JA, Lee S, Ahn JM, Park DW, Kim DH, Kang DH, Song JK, Song JM. Efficacy of 3D transoesophageal echocardiography for transcatheter device closure of atrial septal defect without balloon sizing. Eur Heart J Cardiovasc Imaging. 2018 Jun 1;19(6):684-689. doi: 10.1093/ehjci/jex153. PMID 28633478
- [Background] WINDECKER S, MEIER B. Percutaneous closure of patent foramen ovale, atrial septal defects and the left atrial appendage. Essential Interventional Cardiology (Second Edition): Elsevier; 2008. p. 449-68.